CLINICAL TRIAL: NCT07008443
Title: An Integrated Artificial Intelligence Approach for Predicting Analgesic Time Based on Nalbuphine Versus Morphine as Adjuvants to Bupivacaine in Ultrasound-Guided Supraclavicular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alzahraa Ahmed Abbas (Other)
Responsible Party: Sponsor-Investigator, Alzahraa Ahmed Abbas, Assistant Lecturer of Anesthesia, Damietta Faculty of Medicine, Al-Azhar University, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI-Supraclavicular-Trial-2025
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Regional Anesthesia Block; Upper Limb Surgery
Keywords: Nerve Block Adjuvants Regional Anesthesia; AI Prediction
MeSH Terms: interventions — Bupivacaine; Sodium Chloride; Nalbuphine; Morphine

STUDY DESIGN:
Intervention Model Description: Three-arm parallel design with random assignment to bupivacaine alone, bupivacaine + nalbuphine, or bupivacaine + morphine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and drug preparation were concealed in sealed envelopes. Blinding was maintained for participants, providers, and data analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Bupivacaine + Saline) (Active Comparator): Participants received 25 ml of 0.5% bupivacaine plus 5 ml of normal saline via ultrasound-guided supraclavicular brachial plexus block.
  Interventions: Drug: Bupivacaine + saline
- Nalbuphine Group (Bupivacaine + Nalbuphine) (Experimental): Participants received 25 ml of 0.5% bupivacaine plus nalbuphine at 50 µg/kg via ultrasound-guided supraclavicular brachial plexus block
  Interventions: Drug: Bupivacaine + nalbuphine
- Morphine Group (Bupivacaine + Morphine) (Experimental): Participants received 25 ml of 0.5% bupivacaine plus morphine at 50 µg/kg via ultrasound-guided supraclavicular brachial plexus block.
  Interventions: Drug: Bupivacaine + morphine

INTERVENTIONS:
Drug: Bupivacaine + saline — 25 ml of 0.5% bupivacaine combined with 5 ml of normal saline, administered via ultrasound-guided supraclavicular brachial plexus block as a control intervention
  Arms: Control Group (Bupivacaine + Saline)
Drug: Bupivacaine + nalbuphine — 25 ml of 0.5% bupivacaine combined with nalbuphine at a dose of 50 µg/kg, administered via ultrasound-guided supraclavicular brachial plexus block
  Arms: Nalbuphine Group (Bupivacaine + Nalbuphine)
Drug: Bupivacaine + morphine — 25 ml of 0.5% bupivacaine combined with morphine at a dose of 50 µg/kg, administered via ultrasound-guided supraclavicular brachial plexus block
  Arms: Morphine Group (Bupivacaine + Morphine)

SUMMARY:
This study investigated the effect of adding nalbuphine or morphine to bupivacaine for supraclavicular brachial plexus block in upper limb surgeries. Sixty adult patients were randomized into three groups: control (bupivacaine + saline), nalbuphine, and morphine. The primary objective was to compare the duration of analgesia between the groups. A secondary goal was to assess whether artificial intelligence (AI), specifically the k-nearest neighbor (KNN) algorithm, could predict analgesic duration based on patient clinical and demographic data. The study concluded that both nalbuphine and morphine significantly prolonged analgesic duration and that the AI model showed high predictive accuracy.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind clinical trial was conducted at Al-Zahraa and Damietta University Hospitals to evaluate the effectiveness of nalbuphine and morphine as adjuvants to bupivacaine in ultrasound-guided supraclavicular brachial plexus block. Sixty ASA I-II adult patients scheduled for upper limb surgeries were enrolled and divided equally into three groups. Group C received 0.5% bupivacaine with saline; Group N received bupivacaine with nalbuphine (50 μg/kg); Group M received bupivacaine with morphine (50 μg/kg). The primary outcome was analgesic duration, measured from block performance until the first request for postoperative analgesia. Secondary outcomes included onset and duration of sensory and motor block, total postoperative analgesic consumption, pain scores, and complications.

In parallel, a machine learning model using the K-Nearest Neighbor (KNN) algorithm was developed to predict analgesic duration from demographic and hemodynamic parameters. Exploratory data analysis and clustering methods confirmed the complex relationship between variables. The KNN model demonstrated high predictive accuracy (correlation coefficient ~0.95). The study concluded that both adjuvants extended analgesic duration and that AI models can assist in personalizing analgesic strategies based on patient profiles.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 21-60 years

ASA physical status I or II

Scheduled for elective upper limb surgery below the elbow

Provided written

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Analgesic Duration | From block administration to first request for postoperative analgesia (up to 24 hours)
  Duration of analgesia measured in hours from the time of performing the supraclavicular brachial plexus block until the patient's first request for postoperative pain relief.

SECONDARY OUTCOMES:
Total Postoperative Analgesic Consumption | Within 24 hours postoperatively
  Total amount (in grams) of paracetamol administered as rescue analgesia during the first 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahraa University Hospital, Cairo, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No